CLINICAL TRIAL: NCT02269553
Title: A Pivotal Study of the TMJ NextGeneration(TradeMark) Compared to Occlusal Splint Treatment for Reduction in Nocturnal Bruxism Episodes and Monthly Migraine Episodes in Subjects Diagnosed With Sleep Bruxism
Brief Title: TMJ-1001 Bruxism Run-In/Pivotal Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study redesigned into three separate trials.
Sponsor: TMJ Health (Industry)
Collaborators: Cardiox Corporation (Industry)
Responsible Party: Sponsor
Organization: Cardiox Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMJ-1001
Record Dates: First submitted 2014-10-07; First posted 2014-10-21 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Bruxism
Keywords: Migraine; Headache
MeSH Terms: conditions — Bruxism; Migraine Disorders; Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TMJ NextGeneration(TM) (Active Comparator): The TMJ NextGeneration(TM) device consists of a pair of small, hollow ear inserts. These ear inserts are custom-fit to each subject's ear canals. They are constructed from methacrylate polymers - the same material as has been used in hearing aids. The devices rest in the outer third of the ear canal and have a small retraction post that allows for removal of the device from the ear. The devices conform to the shape of the individuals' ear canals when the jaw is in the open position and permit full passage of sound into each ear. The device is FDA cleared under a 510(k) with an indication of reducing TMD pain.
  Interventions: Device: TMJ(TM) NextGeneration
- Standard Hard TMJD Splint (Active Comparator): The occlusal splint to be used in this study will be a hard, full-arch splint with at least one occlusal contact on each tooth of the opposing arch. Each patient assigned to the occlusal splint treatment group may wear either maxillary or mandibular splints or both, as prescribed by the subject's dentist, during the study. All occlusal splints used in the study will be custom fit to each patient using standard dental processes. All occlusal splints used in the study will be manufactured by Paul O'Neill Dental Lab, Yucaipa , CA, USA using clear ADA approved orthodontic acrylic
  Interventions: Device: Standard Hard TMJD Splint

INTERVENTIONS:
Device: TMJ(TM) NextGeneration — The TMJ NextGeneration(TM) device consists of a pair of small, hollow ear inserts.
  Arms: TMJ NextGeneration(TM)
Device: Standard Hard TMJD Splint — The occlusal splint to be used in this study will be a hard, full-arch splint with at least one occlusal contact on each tooth of the opposing arch.
  Arms: Standard Hard TMJD Splint

SUMMARY:
The study is an open-label, prospective, multi-center, randomized, two treatment parallel, comparison study of the TMJ NextGeneration(TM) and custom-fit occlusal splint in the reduction of nocturnal bruxism episodes and monthly migraine episodes in subjects diagnosed with sleep bruxism and headaches.

DETAILED DESCRIPTION:
The study will be conducted at multiple study centers in the U.S. The study will consist of a screening period lasting up to 5 weeks and a treatment period lasting 8 weeks. Subjects will visit the dental clinic twice during the screening period, at Day 1, and at Weeks 4 and 8 of the study.The study will include a single-center run-in phase during which 12 subjects will be enrolled in order to gain preliminary effectiveness data on the TMJ NextGeneration(TM) device. Following completion of the first 12 subjects, a sample size re-estimation may be conducted in order to verify the initial sample size assumptions of the study. These run-in subjects will not be included in the final analysis of the study. Approximately a total of 153 subjects will be enrolled in the study with subjects allocated 2:1 to the TMJ NextGeneration(TM) and occlusal splint treatment arms, respectively. The study is powered with respect to the dual primary effectiveness endpoints of CFB in bruxism episodes per hour of sleep and CFB in migraine episodes per month.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years of age;
2. Subject has had a diagnosis of sleep bruxism within the past 30 days;
3. Subject is able to read and understand the ICF and has voluntarily provided written informed consent;
4. Subject must have a minimum of 26 remaining teeth;
5. Subject has recorded more than 50% of screening period diary pain VAS scores ≥40;
6. Subject has been medically screened and diagnosed by a physician as having migraines;
7. Subject has been prescribed and is using a triptan as a rescue medication for their migraine episodes;
8. Subject has recorded ≥ 2 self-diagnosed migraine episodes in the screening diary;
9. Subject has an average of ≥ 4 bruxism episodes per hour of sleep based on the screening sleep EMG evaluations;
10. Subject is willing to comply with the usage instructions for the Bruxoff (sleep EMG evaluation) device.
11. Subject is able to open their mouth at least 17 mm to be fitted for the TMJ NextGenerationTM device.
12. Male Subjects are willing to have a clean shaven face on the nights that the Bruxoff device will be used;
13. Subject agrees that when using the Bruxoff device to keep their cellular phone in another room.

Exclusion Criteria:

1. Subjects with any physical or behavioral disorder, which, in the opinion of the Principal Investigator, may interfere with the use of the device or compliance with the study protocol;
2. Subject has any sleep disorder other than bruxism;
3. Subjects who have had direct trauma to the jaw;
4. Subject experiences chronic migraines, > 15 per month;
5. Subject experiences secondary headaches (i.e. Arnold-Chiari syndrome and/or low pressure headaches) in the opinion of the Investigator;
6. Subjects who have used an occlusal appliance to treat TMD within the previous six months;
7. Subjects who have had prior TMJ or ear surgery;
8. Subjects who have a narrow ear canal or impression of the ear canal, which is prolapsed due to an anatomical shift or failure of the ear canal wall structure, or a canal that does not allow for the ear canal second turn to be identified;
9. Subjects with visible or congenital ear deformity as observed on targeted physical exam that does not allow for fitting of the study device;
10. Subjects who have taken a narcotic pain medication in the last seven days prior to Day -7 of the study;
11. Subjects who have a history of ear pain unrelated to TMJ;
12. Subjects who have a history of ear drainage in the past six months;
13. Subjects who have active ear drainage, swelling, or redness as observed on targeted physical exam;
14. Subjects whom the investigator believes may not be an appropriate candidate for an intra-oral splint due to missing or poor quality dentition or untreated pain of dental origin (pulpal pain, pericoronitis of wisdom teeth, or similar conditions);
15. Subjects who, in the opinion of the investigator, cannot be properly fit with their assigned device;
16. Subject has experienced chronic pain (not including migraine pain) associated with sleep bruxism or TMD for more than six months;
17. Subject has a pacemaker.
18. Subject has an allergy to polyethylene, dicumyl peroxide, azodicarbonamide, or ammonia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline (CFB) in bruxism episodes per hour of sleep | Baseline and Week 8
CFB in the number of migraine episodes per month | Baseline and Week 8

SECONDARY OUTCOMES:
CFB in the number of headache episodes per month | Baseline and Week 8
CFB in the in-clinic pain Visual Analogue Scale (VAS) scores | Baseline and Week 8
CFB in the average daily at-home pain VAS scores | Baseline and Week 8
CFB in the morning daily at-home pain VAS scores | Baseline and Week 8
CFB in the evening daily at-home pain VAS scores | Baseline and Week 8

OTHER OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Baseline and Week 8

CONTACTS AND LOCATIONS:
Overall Officials: simon blackburn, CCRA, Study Director — Senior Director, Clinical Affairs